CLINICAL TRIAL: NCT01191268
Title: The Impact of LY2189265 Versus Insulin Glargine in Combination With Insulin Lispro for the Treatment to Target of Type 2 Diabetes Mellitus (AWARD-4: Assessment of Weekly AdministRation of LY2189265 in Diabetes - 4)
Brief Title: A Study in Participants With Type 2 Diabetes Mellitus (AWARD-4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11376; H9X-MC-GBDD (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; dulaglutide; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.5 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Insulin Lispro: dose titration based on blood glucose measures, subcutaneous (SC), thrice daily (after each meal) for 52 weeks
  Interventions: Drug: LY2189265; Drug: Insulin Lispro
- 0.75 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Insulin Lispro: dose titration based on blood glucose measures, subcutaneous (SC), thrice daily (after each meal) for 52 weeks
  Interventions: Drug: LY2189265; Drug: Insulin Lispro
- Insulin Glargine (Active Comparator): Insulin Glargine: dose titration based on blood glucose measures, subcutaneous (SC), once daily for 52 weeks
  Insulin Lispro: dose titration based on blood glucose measures, subcutaneous (SC), thrice daily (after each meal) for 52 weeks
  Interventions: Drug: Insulin Glargine; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Glargine
  Arms: Insulin Glargine
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: 0.75 mg LY2189265; 1.5 mg LY2189265
Drug: Insulin Lispro

SUMMARY:
The purpose of this study is to assess the efficacy and safety of LY2189265 in comparison to Insulin Glargine, both in combination with Insulin Lispro (plus or minus Metformin), in participants with Type 2 Diabetes treated with 1 or 2 injections of insulin.

DETAILED DESCRIPTION:
The term rescue therapy in this trial was defined as therapy for participants who met criteria for persistent severe hyperglycemia and therapy for participants who required new intervention for any other reason. The latter included participants who discontinued study drug due to adverse events, participant decision, or any other reason. For efficacy analyses, participants who received rescue medication were included in the analysis population, but only measurements obtained prior to taking rescue therapy were included in the efficacy analysis. For safety analyses, with the exception of hypoglycemia, all measurements including those obtained after taking rescue therapy were included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently using insulin for at least 3 months with a conventional insulin regimen with or without oral medications
* Glycosylated hemoglobin (HbA1c) greater than or equal to 7% and less than or equal to 11%
* Willing to inject subcutaneous medication
* Willing to monitor blood glucose levels and adjust insulin dose
* Willing to maintain a study diary
* Body mass index (BMI) between 23 and 45 kilograms per square meter (kg/m^2)
* Stable weight for 3 months prior to screening
* Females of child bearing potential must test negative for pregnancy at screening and be willing to use a reliable method of birth control during the study and for 1 month following the last dose of study drug

Exclusion Criteria:

* Type 1 Diabetes
* Previous therapy with glucagon-like peptide 1 (GLP-1) agonists within 3 months prior to screening
* 1 or more episodes of ketoacidosis within 6 months prior to screening
* Have been treated with prescription or over the counter medication to promote weight loss within 3 months prior to screening
* Estimated glomerular filtration rate (eGFR) less than or equal to 30 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2) at screening
* Taking steroids for greater than 14 days except for topical, eye, nasal, or inhaled
* History of heart failure, New York Heart Classification III or IV within 2 months prior to screening
* Gastrointestinal (GI) problems such as diabetic gastroparesis or bariatric surgery (stomach stapling) or chronically taking medications that directly affect GI motility
* Acute or chronic hepatitis or pancreatitis
* Self or family history of 2A or type 2B multiple endocrine neoplasia or medullary C-Cell hyperplasia
* Serum calcitonin greater than or equal to 20 picograms per milliliter (pcg/mL) at screening
* Organ transplant except cornea
* Significant active autoimmune disease such as Lupus or Rheumatoid Arthritis
* History of or active malignancy except skin or in situ cervical or prostate cancer within the last 5 years
* Known drug or alcohol abuse
* Have enrolled in another clinical trial within the last 30 days
* Have previously signed an informed consent or participated in a LY2189265 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (101):
- United States (36):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Haven, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paducah, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waltham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cipolletti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salta
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonheiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belém
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Westminster, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gatineau, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Denmark (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hillerød
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Koege
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolding
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nikaias - Piraeus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyöngyös
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miskolc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagykanizsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pápa
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Culiacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Radzymin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yabucoa
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Samara
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karlstad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yongkang District

REFERENCES:
- [Derived] Pantalone KM, Patel H, Yu M, Fernandez Lando L. Dulaglutide 1.5 mg as an add-on option for patients uncontrolled on insulin: Subgroup analysis by age, duration of diabetes and baseline glycated haemoglobin concentration. Diabetes Obes Metab. 2018 Jun;20(6):1461-1469. doi: 10.1111/dom.13252. Epub 2018 Mar 23. PMID 29430801
- [Derived] Boustani MA, Pittman I 4th, Yu M, Thieu VT, Varnado OJ, Juneja R. Similar efficacy and safety of once-weekly dulaglutide in patients with type 2 diabetes aged >/=65 and <65 years. Diabetes Obes Metab. 2016 Aug;18(8):820-8. doi: 10.1111/dom.12687. Epub 2016 Jun 7. PMID 27161178
- [Derived] Yu M, Van Brunt K, Varnado OJ, Boye KS. Patient-reported outcome results in patients with type 2 diabetes treated with once-weekly dulaglutide: data from the AWARD phase III clinical trial programme. Diabetes Obes Metab. 2016 Apr;18(4):419-24. doi: 10.1111/dom.12624. Epub 2016 Feb 4. PMID 26691396
- [Derived] Blonde L, Jendle J, Gross J, Woo V, Jiang H, Fahrbach JL, Milicevic Z. Once-weekly dulaglutide versus bedtime insulin glargine, both in combination with prandial insulin lispro, in patients with type 2 diabetes (AWARD-4): a randomised, open-label, phase 3, non-inferiority study. Lancet. 2015 May 23;385(9982):2057-66. doi: 10.1016/S0140-6736(15)60936-9. PMID 26009229

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Started | 295 | 293 | 296
Received at Least One Dose of Study Drug | 295 | 293 | 296
Completed | 237 | 238 | 244
Not Completed | 58 | 55 | 52
Not completed — Withdrawal by Subject | 19 | 25 | 21
Not completed — Adverse Event | 21 | 13 | 8
Not completed — Physician Decision | 6 | 8 | 9
Not completed — Lost to Follow-up | 8 | 5 | 9
Not completed — Entry Criteria Not Met | 3 | 1 | 1
Not completed — Death | 0 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Sponsor Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least 1 dose of LY2189265 or Insulin Glargine.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine | Total
Number analyzed (Participants) | 295 | 293 | 296 | 884
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.88 (9.55) | 59.31 (8.98) | 59.90 (9.08) | 59.36 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 145 | 131 | 411
  Male | 160 | 148 | 165 | 473
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102 | 101 | 100 | 303
  Not Hispanic or Latino | 193 | 192 | 196 | 581
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 13 | 17 | 46
  Asian | 9 | 12 | 14 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 32 | 27 | 26 | 85
  White | 231 | 235 | 231 | 697
  More than one race | 7 | 6 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 103 | 95 | 96 | 294
  Taiwan | 8 | 9 | 9 | 26
  Greece | 8 | 7 | 8 | 23
  Spain | 8 | 10 | 9 | 27
  Russian Federation | 6 | 8 | 9 | 23
  Hungary | 19 | 19 | 19 | 57
  Mexico | 19 | 19 | 17 | 55
  Canada | 9 | 8 | 9 | 26
  Puerto Rico | 13 | 20 | 18 | 51
  Argentina | 26 | 27 | 28 | 81
  Poland | 13 | 13 | 14 | 40
  Brazil | 33 | 30 | 32 | 95
  Belgium | 5 | 5 | 4 | 14
  Denmark | 4 | 4 | 4 | 12
  Australia | 10 | 8 | 8 | 26
  Sweden | 11 | 11 | 12 | 34
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 91.00 (18.24) | 91.69 (18.03) | 90.75 (18.87) | 91.14 (18.37)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 31.99 (5.11) | 33.08 (5.15) | 32.41 (5.33) | 32.49 (5.21)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.46 (1.08) | 8.40 (1.03) | 8.53 (1.03) | 8.46 (1.05)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 12.80 (7.19) | 12.43 (6.92) | 12.96 (6.80) | 12.73 (6.97)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 26-week Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, baseline metformin, and baseline HbA1c.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable HbA1c data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 273 | 275 | 276
percentage of glycosylated hemoglobin | -1.64 (0.07) | -1.59 (0.07) | -1.41 (0.07)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; The study was designed to enroll 837 randomized participants (279 per treatment arm) with 90% power to detect non-inferiority of 1.5 mg LY2189265 versus Insulin Glargine on HbA1c change from baseline at the 26-week primary endpoint with a margin of 0.4%, a standard deviation of 1.3%, and a 1-sided alpha of 0.025 assuming no true difference between treatments. This corresponds to 248 participants per arm, with an assumed drop-out rate of 11%; Test type: Non-Inferiority or Equivalence — If the upper limit of the 95% Confidence Interval (CI) of 1.5 mg LY2189265 versus Insulin Glargine was below 0.4%, 1.5 mg LY2189265 was declared non-inferior to Insulin Glargine; p < 0.001, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.22, 95% CI 2-sided [-0.38 to -0.07]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — If the 1-sided adjusted p-value was below 0.025, then 0.75 mg LY2189265 was declared non-inferior to Insulin Glargine; p < 0.001, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.17, 95% CI 2-sided [-0.33 to -0.02]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p = 0.005, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.22, 95% CI 2-sided [-0.38 to -0.07]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p = 0.015, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.17, 95% CI 2-sided [-0.33 to -0.02]

2. Secondary Outcome: Change From Baseline to 52-week Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: as for outcome 1
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 273 | 275 | 276
percentage of glycosylated hemoglobin | -1.48 (0.08) | -1.42 (0.08) | -1.23 (0.08)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.25, 95% CI 2-sided [-0.42 to -0.07]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — If the 1-sided adjusted p-value was below 0.025, then 0.75 mg LY2189265 was declared non-inferior to Insulin Glargine; p < 0.001, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.19, 95% CI 2-sided [-0.37 to -0.02]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p = 0.005, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.25, 95% CI 2-sided [-0.42 to -0.07]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Superiority analysis; Test type: Superiority or Other; p = 0.014, ANCOVA — Family-wise Type I error rate was controlled by applying tree-gatekeeping strategy; LS Mean Difference = -0.19, 95% CI 2-sided [-0.37 to -0.02]

3. Secondary Outcome: Percentage of Participants Attaining Glycosylated Hemoglobin (HbA1c) Less Than 7% and Less Than or Equal to 6.5% at Weeks 26 and 52
Description: The percentage of participants achieving HbA1c level less than 7.0% and less than or equal to 6.5% was analyzed with a repeated logistic regression model (generalized estimating equation model) with baseline HbA1c, baseline metformin, country, and treatment as factors included in the model.
Time Frame: 26 weeks and 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 275 | 277 | 280
percentage of participants
  HbA1c less than 7.0%, 26 weeks | 67.6 | 69.0 | 56.8
  HbA1c less than 7.0%, 52 weeks | 58.5 | 56.3 | 49.3
  HbA1c less than or equal to 6.5%, 26 weeks | 48.0 | 43.0 | 37.5
  HbA1c less than or equal to 6.5%, 52 weeks | 36.7 | 34.7 | 30.4
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.014, Regression, Logistic — Treatment comparison for HbA1c less than 7.0% at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.010, Regression, Logistic — Treatment comparison for HbA1c less than 7.0% at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.027, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 26 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.384, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 26 weeks
Statistical Analysis 5: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.05, Regression, Logistic — Treatment comparison for HbA1c less than 7% at 52 weeks
Statistical Analysis 6: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.250, Regression, Logistic — Treatment comparison for HbA1c less than 7% at 52 weeks
Statistical Analysis 7: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.272, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 52 weeks
Statistical Analysis 8: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.623, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5% at 52 weeks

4. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Percentage of Participants Achieving Glycosylated Hemoglobin (HbA1c) Less Than 7% Without Nocturnal or Severe Hypoglycemia
Description: The percentage of participants achieving HbA1c less than 7.0% without nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking) or severe (episodes requiring the assistance of another person to actively administer resuscitative actions) hypoglycemia was analyzed with a repeated logistic regression model (generalized estimating equation model) with baseline HbA1c, baseline metformin, country, and treatment as factors included in the model.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 275 | 277 | 280
percentage of participants
  26 weeks | 53.8 | 54.5 | 28.2
  52 weeks | 44.0 | 44.0 | 26.8
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 26 weeks
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 26 weeks
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 52 weeks
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison at 52 weeks

5. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Blood Glucose Values From the 8-point Self-monitored Plasma Glucose (SMPG) Profiles
Description: The self-monitored plasma glucose (SMPG) data were collected at the following 8 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening meal; 2 hours post-evening meal; bedtime; and 3AM or 5 hours after bedtime. The mean of the 8 time points (Daily Mean) was also calculated. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, metformin, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable SMPG data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)]
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
millimoles per liter (mmol/L)]
  Pre-morning meal, 26 weeks (n=228, 231, 232) | -0.36 (0.14) | -0.06 (0.14) | -2.01 (0.14)
  Post-morning meal, 26 weeks (n=220, 227, 229) | -3.70 (0.19) | -3.29 (0.19) | -4.03 (0.18)
  Pre-midday meal, 26 weeks (n=227, 231, 233) | -2.80 (0.16) | -2.38 (0.16) | -2.65 (0.16)
  Post-midday meal, 26 weeks (n=219, 227, 228) | -4.51 (0.17) | -4.53 (0.17) | -3.70 (0.17)
  Pre-evening meal, 26 weeks (n=226, 231, 232) | -3.24 (0.16) | -3.06 (0.16) | -2.74 (0.16)
  Post-evening meal, 26 weeks (n=220, 228, 227) | -4.61 (0.17) | -4.54 (0.17) | -3.90 (0.17)
  Bedtime, 26 weeks (n=220, 221, 226) | -4.00 (0.17) | -3.89 (0.17) | -3.40 (0.17)
  After bedtime, 26 weeks (n=208, 216, 208) | -1.48 (0.15) | -1.50 (0.15) | -1.96 (0.15)
  Daily Mean, 26 weeks (n=202, 206, 199) | -3.17 (0.12) | -2.97 (0.12) | -3.10 (0.12)
  Pre-morning meal, 52 weeks (n=207, 213, 218) | 0.03 (0.16) | 0.05 (0.15) | -2.02 (0.15)
  Post-morning meal, 52 weeks (n=200, 211, 211) | -3.38 (0.19) | -3.23 (0.19) | -3.76 (0.19)
  Pre-midday meal, 52 weeks (n=207, 213, 218) | -2.53 (0.14) | -2.52 (0.14) | -2.63 (0.14)
  Post-midday meal, 52 weeks (n=202, 210, 212) | -4.33 (0.18) | -4.29 (0.18) | -3.83 (0.18)
  Pre-evening meal, 52 weeks (n=207, 214, 217) | 3.00 (0.16) | -3.07 (0.16) | -2.67 (0.16)
  Post-evening meal, 52 weeks (n=200, 210, 212) | -4.22 (0.17) | -4.54 (0.17) | -3.71 (0.16)
  Bedtime, 52 weeks (n=195, 205, 213) | -3.62 (0.17) | -3.96 (0.17) | -3.27 (0.17)
  After bedtime, 52 weeks (n=192, 192 197) | -1.17 (0.15) | -1.36 (0.15) | -1.80 (0.15)
  Daily Mean, 52 weeks (n=182, 185, 189) | -2.84 (0.12) | -2.95 (0.12) | -2.97 (0.12)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.628, Mixed Models Analysis — Treatment comparison of Daily Mean values at 26 weeks; LS Mean Difference = -0.07, 95% CI 2-sided [-0.35 to 0.21]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.368, Mixed Models Analysis — Treatment comparison of Daily Mean values at 26 weeks; LS Mean Difference = 0.13, 95% CI 2-sided [-0.15 to 0.41]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.370, Mixed Models Analysis — Treatment comparison of Daily Mean values at 52 weeks; LS Mean Difference = 0.13, 95% CI 2-sided [-0.16 to 0.42]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p = 0.879, Mixed Models Analysis — Treatment comparison of Daily Mean values at 52 weeks; LS Mean Difference = 0.02, 95% CI 2-sided [-0.26 to 0.30]

6. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Fasting Serum Glucose
Description: Fasting serum glucose was measured by the central laboratory. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, metformin use, and treatment-by-visit interaction as fixed effects and baseline fasting blood glucose as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable fasting blood glucose data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 292 | 294
millimoles per liter (mmol/L)
  26 weeks (n=253, 256, 255) | -0.27 (0.20) | 0.22 (0.20) | -1.58 (0.20)
  52 weeks (n=237, 238, 246) | 0.08 (0.22) | 0.41 (0.22) | -1.01 (0.22)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks; LS Mean Difference = 1.31, 95% CI 2-sided [0.83 to 1.79]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks; LS Mean Difference = 1.80, 95% CI 2-sided [1.32 to 2.28]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 52 weeks; LS Mean Difference = 1.09, 95% CI 2-sided [0.55 to 1.64]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 52 weeks; LS Mean Difference = 1.42, 95% CI 2-sided [0.88 to 1.96]

7. Secondary Outcome: Total Daily Insulin Dose Overall and by Components (Insulin Lispro and Insulin Glargine)
Description: Total daily insulin (TDI) dose was reported at baseline, 26 weeks, and 52 weeks. Daily Insulin Lispro and Insulin Glargine doses were reported at 26 and 52 weeks.
Time Frame: Baseline and 26 weeks and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
units
  TDI, Baseline | 55.20 (32.17) | 59.11 (38.12) | 53.93 (30.67)
  TDI, 26 weeks (n=244, 251, 254) | 93.24 (78.02) | 96.69 (62.13) | 132.00 (79.01)
  TDI, 52 weeks (n=224, 227, 238) | 88.15 (62.95) | 95.00 (67.62) | 133.19 (80.75)
  Insulin Lispro, 26 weeks (n=244, 251, 254) | 93.24 (78.02) | 96.69 (62.13) | 67.79 (44.59)
  Insulin Lispro, 52 weeks (n=224, 227, 238) | 88.15 (62.95) | 95.00 (67.62) | 69.12 (49.07)
  Insulin Glargine, 26 weeks (n=244, 251, 254) | NA (NA) — Participants in this treatment arm were not exposed to Insulin Glargine. | NA (NA) — Participants in this treatment arm were not exposed to Insulin Glargine. | 64.48 (40.23)
  Insulin Glargine, 52 weeks (n=224, 227, 238) | NA (NA) — Participants in this treatment arm were not exposed to Insulin Glargine. | NA (NA) — Participants in this treatment arm were not exposed to Insulin Glargine. | 64.07 (38.60)

8. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Body Weight
Description: Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country, treatment, and metformin use as fixed effects and baseline body weight as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable body weight data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 286 | 289 | 294
kilograms (kg)
  26 weeks | -0.87 (0.27) | 0.18 (0.27) | 2.33 (0.27)
  52 weeks | -0.35 (0.34) | 0.86 (0.33) | 2.89 (0.33)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 26 weeks; LS Mean Difference = -3.20, 95% CI 2-sided [-3.81 to -2.59]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 26 weeks; LS Mean Difference = -2.15, 95% CI 2-sided [-2.76 to -1.54]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 52 weeks; LS Mean Difference = -3.23, 95% CI 2-sided [-3.99 to -2.48]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison at 52 weeks; LS Mean Difference = -2.03, 95% CI 2-sided [-2.78 to -1.27]

9. Secondary Outcome: Body Weight at Baseline, 52 Weeks, and 4 Weeks After Last Dose
Time Frame: Baseline and 52 weeks and 4 weeks after last dose
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable body weight data.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
kilograms (kg)
  Baseline | 91.00 (18.24) | 91.69 (18.03) | 90.75 (18.87)
  52 weeks (n=290, 290, 295) | 91.58 (19.06) | 93.21 (19.23) | 94.14 (19.72)
  4 weeks after last dose (n=259, 260, 253) | 91.69 (18.60) | 93.14 (19.20) | 94.27 (20.13)

10. Secondary Outcome: Change From Baseline to 26 Weeks, 52 Weeks, and 4 Weeks After Last Dose in Body Mass Index (BMI)
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, metformin use, and treatment-by-visit interaction as fixed effects and baseline BMI as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable BMI data.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
kilograms per meter squared (kg/m^2)
  26 weeks (n=248, 251, 250) | -0.20 (0.09) | 0.21 (0.09) | 1.01 (0.09)
  52 weeks (n=225, 224, 232) | 0.09 (0.11) | 0.57 (0.11) | 1.33 (0.11)
  4 weeks after last dose | NA (NA) — Data from 4 weeks after last dose was not analyzed for this outcome. | NA (NA) — Data from 4 weeks after last dose was not analyzed for this outcome. | NA (NA) — Data from 4 weeks after last dose was not analyzed for this outcome.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks; LS Mean Difference = -1.20, 95% CI 2-sided [-1.44 to -0.96]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks; LS Mean Difference = -0.79, 95% CI 2-sided [-1.03 to -0.55]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 52 weeks; LS Mean Difference = -1.24, 95% CI 2-sided [-1.55 to -0.94]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 52 weeks; LS Mean Difference = -0.76, 95% CI 2-sided [-1.06 to -0.46]

11. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the EQ-5D
Description: The EQ-5D questionnaire is a generic, multidimensional, health-related, quality-of-life instrument. It consists of 2 parts: the first part assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that have 3 possible levels of response (no problem, some problem, or extreme problem). These dimensions are converted into a weighted health-state Index Score. The EQ-5D United Kingdom (UK) score ranges from -0.59 to 1.0, where a score of 1.0 indicates perfect health and negative values are valued as worse than dead. The second part consists of a visual analog scale (VAS) on which the participants rated their perceived health state on that day from 0 (worst imaginable health state) to 100 (best imaginable health). Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) adjusted by treatment, country, metformin use, and baseline.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable EQ-5D data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
units on a scale
  EQ-5D UK, 26 weeks (n=272, 271, 274) | -0.03 (0.01) | -0.03 (0.01) | -0.03 (0.01)
  EQ-5D UK, 52 weeks (n=274, 274, 281) | -0.04 (0.01) | -0.04 (0.01) | -0.03 (0.01)
  VAS, 26 weeks (n=278, 275, 275) | -1.69 (1.00) | -2.30 (1.00) | -0.60 (1.00)
  VAS, 52 weeks (n=279, 278, 282) | -0.46 (1.01) | -2.54 (1.02) | -0.18 (1.01)

12. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Impact of Weight on Activities of Daily Living (IW-ADL)
Description: The Impact of Weight on Activities of Daily Living questionnaire (renamed the Ability to Perform Physical Activities of Daily Living Questionnaire [APPADL]) contains 7 items that assess how difficult it is for participants to engage in certain activities considered to be integral to normal daily life, such as walking, standing and climbing stairs. Items are scored on a 5-point numeric rating scale where 5 = "not at all difficult" and 1 = "unable to do". The individual scores from all 7 items are summed and a single total score is calculated and may range between 7 and 35. A higher score indicates better ability to perform activities of daily living. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country, treatment, and metformin use as fixed effects and baseline score as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable APPADL data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 293 | 290 | 294
units on a scale
  26 weeks (n=274, 270, 270) | -0.50 (0.30) | -0.60 (0.31) | -0.93 (0.31)
  52 weeks (n=277, 275, 279) | -0.50 (0.33) | -1.05 (0.33) | -1.28 (0.33)

13. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Impact of Weight on Self-Perception (IW-SP)
Description: The Impact of Weight on Self-Perception (IW-SP) questionnaire contains 3 items that assess how often the participants' body weight affects how happy they are with their appearance and how often they feel self-conscious when out in public. Items are scored on a 5-point numeric rating scale where 5 = never and 1 = always. A single total score is calculated by summing the scores for all 3 items. Total score ranges between 3 and 15, where a higher score is indicative of better self-perception. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country, treatment, and metformin use as fixed effects and baseline score as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable IW-SP data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 293 | 291 | 295
units on a scale
  26 weeks (n=277, 274, 274) | 0.60 (0.17) | 0.34 (0.17) | 0.18 (0.17)
  52 weeks (n=278, 277, 281) | 0.86 (0.16) | 0.22 (0.16) | 0.06 (0.16)

14. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in the Low Blood Sugar Survey (LBSS)
Description: The Low Blood Sugar Survey (LBSS) contains 33 items comprised of 2 subscales (behavior and worry), each of which is rated on a 5-point numeric rating scale from 0 (never) to 4 (almost always). It captures behavioral changes associated with the concerns and experiences of hypoglycemia and the degree to which participants are worried about certain aspects associated with hypoglycemia during the previous 4 weeks. The behavior (or avoidance) subscale has 15 items, and the worry (or affect) subscale has 18 items. Subscale scores are calculated by summing participant responses to items (behavior range 0-60; worry range 0-72). A total score is calculated as the sum of both subscales (range 0-132). Higher scores indicate greater negative impact on subscales and total score. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country, treatment and metformin use as fixed effects and baseline score as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable LBSS data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 293 | 292 | 296
units on a scale
  26 weeks (n=251, 256, 250) | 3.75 (1.31) | 2.91 (1.29) | 2.83 (1.30)
  52 weeks (n=234, 238, 244) | 2.51 (1.25) | 0.92 (1.23) | 2.38 (1.23)

15. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Pancreatic Enzymes
Description: Amylase (total and pancreas-derived [PD]) and lipase concentrations were measured.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable pancreatic enzyme data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units per liter (U/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
units per liter (U/L)
  Amylase (total), 26 weeks (n=284, 282, 287) | 5.00 [-2.00 to 15.00] | 4.00 [-1.00 to 10.00] | 1.00 [-4.00 to 8.00]
  Amylase (total), 52 weeks (n=284, 283, 287) | 2.00 [-3.00 to 12.00] | 2.00 [-4.00 to 9.00] | 0.00 [-7.00 to 6.00]
  Amylase (PD), 26 weeks (n=284, 282, 287) | 4.00 [0.00 to 10.00] | 2.50 [0.00 to 7.00] | 1.00 [-2.00 to 4.00]
  Amylase (PD), 52 weeks (n=284, 283, 287) | 3.00 [-2.00 to 9.00] | 2.00 [-2.00 to 5.00] | 0.00 [-3.00 to 3.00]
  Lipase, 26 weeks (n=284, 282, 287) | 7.00 [0.00 to 17.00] | 4.00 [-3.00 to 12.00] | -2.00 [-8.00 to 3.00]
  Lipase, 52 weeks (n=284, 283, 287) | 6.00 [-1.00 to 16.50] | 3.00 [-3.00 to 11.00] | -2.00 [-9.00 to 4.00]

16. Secondary Outcome: Pancreatic Enzymes at Baseline, 52 Weeks, and 4 Weeks After Last Dose
Description: Amylase (total and pancreas-derived [PD]) and lipase concentrations were measured at baseline and at 4 weeks after last dose (ALD).
Time Frame: Baseline and 52 weeks and 4 weeks after last dose
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable pancreatic enzyme data.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
units per liter (U/L)
  Amylase (total), Baseline | 61.21 (27.89) | 58.59 (23.19) | 61.18 (26.69)
  Amylase (total), 52 weeks (n=284, 283, 287) | 66.08 (30.29) | 60.97 (25.78) | 61.93 (27.12)
  Amylase (total), 4 weeks ALD (n=251, 259, 251) | 61.69 (28.06) | 59.21 (30.32) | 62.13 (26.11)
  Amylase (PD), Baseline | 26.56 (14.51) | 25.10 (13.48) | 26.43 (15.94)
  Amylase (PD), 52 weeks (n=284, 283, 287) | 31.38 (18.15) | 27.86 (17.14) | 26.91 (17.64)
  Amylase (PD), 4 weeks ALD (n=251, 260, 251) | 27.50 (15.49) | 25.77 (13.78) | 26.84 (15.44)
  Lipase, Baseline | 41.42 (34.19) | 41.08 (32.80) | 43.20 (37.35)
  Lipase, 52 weeks (n=284, 283, 287) | 50.57 (35.65) | 45.34 (31.23) | 39.39 (27.51)
  Lipase, 4 weeks ALD (n=252, 260, 251) | 44.19 (36.92) | 41.86 (25.22) | 43.02 (35.75)

17. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Serum Calcitonin
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable serum calcitonin data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing
Measure: Median (Inter-Quartile Range); unit: picogram per milliliter (pcg/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 294 | 293 | 296
picogram per milliliter (pcg/mL)
  26 weeks (n=283, 282, 285) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  52 weeks (n=283, 283, 285) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

18. Secondary Outcome: Serum Calcitonin at Baseline, 52 Weeks, and 4 Weeks After Last Dose
Time Frame: Baseline and 52 weeks and 4 weeks after last dose
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable serum calcitonin data.
Measure: Mean (Standard Deviation); unit: picomole per liter
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 294 | 293 | 296
picomole per liter
  Baseline | 0.75 (0.78) | 0.73 (0.77) | 0.78 (0.88)
  52 weeks (n=284, 283, 285) | 0.79 (0.89) | 0.78 (0.90) | 0.80 (0.89)
  4 weeks after last dose (n=245, 254, 246) | 0.76 (0.87) | 0.73 (0.72) | 0.87 (0.95)

19. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Blood Pressure
Description: Seated systolic blood pressure (SBP) and seated diastolic blood pressure (DBP) were measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, metformin use, and treatment-by-visit interaction as fixed effects and baseline blood pressure as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: milliliters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
milliliters of mercury (mmHg)
  SBP, 26 weeks (n=255, 261, 258) | -0.97 (0.88) | -0.65 (0.87) | 2.23 (0.88)
  SBP, 52 weeks (n=239, 240, 246) | -0.26 (0.94) | 1.04 (0.93) | 1.98 (0.92)
  DBP, 26 weeks (n=255, 261, 258) | 0.02 (0.56) | -0.08 (0.56) | -0.23 (0.56)
  DBP, 52 weeks (n=239, 240, 246) | -0.01 (0.57) | 0.15 (0.57) | -0.34 (0.56)

20. Secondary Outcome: Blood Pressure at Baseline, 52 Weeks, and 4 Weeks After Last Dose
Description: Seated systolic blood pressure (SBP) and seated diastolic blood pressure (DBP) were measured.
Time Frame: Baseline and 52 weeks and 4 weeks after last dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: milliliters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
milliliters of mercury (mmHg)
  SBP, Baseline | 133.26 (16.56) | 134.03 (15.87) | 133.26 (16.97)
  SBP, 52 weeks (n=290, 290, 295) | 132.67 (15.40) | 134.31 (16.41) | 134.90 (16.25)
  SBP, 4 weeks after last dose (n=260, 260, 255) | 133.77 (16.80) | 134.72 (16.50) | 132.75 (16.01)
  DBP, Baseline | 77.33 (9.73) | 77.57 (9.00) | 77.18 (10.41)
  DBP, 52 weeks (n=290, 290, 295) | 77.33 (9.63) | 77.59 (9.74) | 77.07 (9.92)
  DBP, 4 weeks after last dose (n=260, 260, 255) | 76.58 (10.06) | 77.04 (9.60) | 76.94 (9.10)

21. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Pulse Rate
Description: Seated pulse rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, metformin use, and treatment-by-visit interaction as fixed effects and baseline as a covariate
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable seated pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
beats per minute (bpm)
  26 weeks (n=255, 261, 258) | 2.84 (0.57) | 2.79 (0.56) | 0.90 (0.56)
  52 weeks (n=239, 240, 246) | 2.38 (0.57) | 2.27 (0.57) | 0.93 (0.57)

22. Secondary Outcome: Pulse Rate at Baseline, 52 Weeks, and 4 Weeks After Last Dose
Description: Seated pulse rate was measured.
Time Frame: Baseline and 52 weeks and 4 weeks after last dose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
beats per minute (bpm)
  Baseline | 75.26 (11.03) | 75.08 (11.10) | 74.54 (10.50)
  52 weeks (n=290, 290, 295) | 78.30 (11.01) | 77.83 (10.90) | 76.02 (11.43)
  4 weeks after last dose (n=260, 260, 255) | 74.52 (11.09) | 74.99 (11.98) | 75.27 (11.17)

23. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, metformin use, and treatment-by-visit interaction as fixed effects and baseline value as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable ECG QTcF or PR Interval data.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
milliseconds (msec)
  QTcF interval, 26 weeks (n=241, 242, 236) | 0.29 (1.13) | 0.30 (1.12) | 1.59 (1.13)
  QTcF interval, 52 weeks (n= 222, 221, 221) | 1.89 (1.13) | 1.48 (1.13) | 1.80 (1.14)
  PR interval, 26 weeks (n=238, 243, 236) | 0.82 (0.95) | -1.75 (0.94) | -1.13 (0.95)
  PR interval, 52 weeks (n=220, 222, 221) | 0.85 (1.00) | 0.05 (0.99) | -0.43 (1.00)

24. Secondary Outcome: Change From Baseline to 26 and 52 Weeks in Electrocardiogram Parameters, Heart Rate
Description: Electrocardiogram (ECG) heart rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, metformin use, and treatment-by-visit interaction as fixed effects and baseline value as a covariate.
Time Frame: Baseline, 26 weeks, and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine with evaluable ECG heart rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 294 | 293 | 296
beats per minute (bpm)
  26 weeks (n=244, 246, 243) | 3.95 (0.65) | 4.18 (0.65) | 1.37 (0.65)
  52 weeks (n=230, 226, 230) | 3.02 (0.67) | 3.83 (0.67) | 1.03 (0.67)

25. Secondary Outcome: Number of Events of Adjudicated Pancreatitis up to 26 Weeks, 52 Weeks, and 4 Weeks After Last Dose
Description: The number of adjudicated (by an independent Clinical Endpoint Committee [CEC]) pancreatic events is summarized at 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: events
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
events
  26 weeks | NA — Data from 26 weeks was not analyzed for this outcome. | NA — Data from 26 weeks was not analyzed for this outcome. | NA — Data from 26 weeks was not analyzed for this outcome.
  52 weeks | 0 | 0 | 0
  4 weeks after last dose | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome.

26. Secondary Outcome: Number of Participants With Self-reported Hypoglycemic Events up to 26 Weeks, 52 Weeks, and 4 Weeks After Last Dose
Description: Hypoglycemic events (HE) were classified as severe (episodes requiring the assistance of another person to actively administer resuscitative actions and had a plasma glucose [PG] of ≤ 70 milligrams per deciliter [mg/dL]), documented symptomatic (any time a participant felt that he/she was experiencing symptoms and/or signs associated with hypoglycemia and had a PG of ≤ 70 mg/dL), or asymptomatic (events not accompanied by typical symptoms of hypoglycemia but with a measured PG of ≤ 70 mg/dL). The number of participants with self-reported hypoglycemic events is summarized cumulatively. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine. Only pre-rescue measurements were used.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
participants
  Severe HE, 26 weeks | 4 | 5 | 9
  Severe HE, 52 weeks | 8 | 7 | 14
  Severe HE, 4 weeks after last dose | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome.
  Documented Symptomatic HE, 26 weeks | 228 | 242 | 243
  Documented Symptomatic HE, 52 weeks | 235 | 250 | 247
  Documented Symptomatic HE, 4 weeks after last dose | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome.
  Asymptomatic HE, 26 weeks | 174 | 179 | 198
  Asymptomatic HE, 52 weeks | 191 | 196 | 207
  Asymptomatic HE, 4 weeks after last dose | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome.
  Total HE, 26 weeks | 250 | 258 | 264
  Total HE, 52 weeks | 252 | 263 | 266
  Total HE, 4 weeks after last dose | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome. | NA — Data from 4 weeks after last dose was not analyzed for this outcome.

27. Secondary Outcome: Rate of Self-reported Hypoglycemic Events up to 52 Weeks
Description: Hypoglycemic events (HE) were classified as severe (episodes requiring the assistance of another person to actively administer resuscitative actions and had a plasma glucose [PG] of ≤ 70 milligrams per deciliter [mg/dL]), documented symptomatic (any time a participant felt that he/she was experiencing symptoms and/or signs associated with hypoglycemia and had a PG of ≤ 70 mg/dL), or asymptomatic (events not accompanied by typical symptoms of hypoglycemia but with a measured PG of ≤ 70 mg/dL). The 1-year adjusted rate of hypoglycemic events is summarized cumulatively at 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
events per participant per year
  Severe HE | 0.03 (0.19) | 0.05 (0.50) | 0.08 (0.43)
  Documented Symptomatic HE | 30.98 (39.64) | 35.03 (44.94) | 39.90 (50.92)
  Asymptomatic HE | 9.55 (19.52) | 11.56 (24.69) | 14.20 (23.19)
  Total HE | 41.52 (46.51) | 47.42 (54.39) | 55.93 (59.46)

28. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events up to 52 Weeks
Description: Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular AEs to be adjudicated include myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
participants
  Any cardiovascular event | 5 | 6 | 12
  Any fatal cardiovascular event | 0 | 0 | 2
  Any non-fatal cardiovascular event | 5 | 6 | 11

29. Secondary Outcome: Number of Participants With Treatment Emergent LY2189265 Antibodies up to 26 Weeks, 52 Weeks, and 4 Weeks After Last Dose
Description: A participant was considered to have treatment emergent LY2189265 anti-drug antibodies (ADA) if the participant had at least one titer that was treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline through 4 weeks after last dose
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 ADA data.
Measure: Number; unit: participants
Groups:
- 1.5 mg or 0.75 mg LY2189265: LY2189265 (Dulaglutide): 1.5 milligrams (mg) or 0.75 mg , subcutaneous (SC), once weekly for 52 weeks
  Insulin Lispro: dose titration based on blood glucose measures, subcutaneous (SC), thrice daily (after each meal) for 52 weeks
Arm/Group | 1.5 mg or 0.75 mg LY2189265
Number analyzed (Participants) | 562
participants
  26 weeks | NA — Data from 26 weeks was not analyzed for this outcome.
  52 weeks | NA — Data from 52 weeks was not analyzed for this outcome.
  4 weeks after last dose | 9

30. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events up to 26 Weeks, 52 Weeks, and 4 Weeks After Last Dose
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with one or more TEAE is summarized cumulatively at 26 weeks, 52 weeks, and 4 weeks after last dose. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks, 52 weeks, and 4 weeks after last dose
Population: Participants who were randomized and received at least one dose of LY2189265 or Insulin Glargine.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Number analyzed (Participants) | 295 | 293 | 296
participants
  26 weeks | 203 | 216 | 178
  52 weeks | 217 | 230 | 206
  4 weeks after last dose | 223 | 235 | 211

ADVERSE EVENTS:
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 27/295 | 46/293 | 53/296
Other Adverse Events (participants affected / at risk) | 219/295 | 232/293 | 203/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg LY2189265 (N=295) | 0.75 mg LY2189265 (N=293) | Insulin Glargine (N=296)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhagic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block third degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Event resulted in death
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary atherosclerosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Decompensated heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fibrillation ventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Heart block third degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Infarct myocardial (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Non st segment elevation myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Non stemi (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Unstable angina (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Event resulted in death
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Retinal hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal herniation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis noninfectious (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoidal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paralytic ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain exertional (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ancylostomiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Cellulitis of foot (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of leg (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gangrenous appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hookworm infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected toe (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pleurisy viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (5) | 1 (1) — One event resulted in one death in 0.75 mg LY2189265 arm
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) — One event resulted in one death in 1.5 mg LY2189265 arm
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus aureus septicemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Supraglottitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Falling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured ribs (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fractured sternum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Knee fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Leg injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture l1 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Quadriceps tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Torn muscle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 8 (17) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (7) | 7 (16) | 12 (20)
Hypoglycemic episode (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis aggravated (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/160 (0) | 1/148 (1) | 0/165 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumboischialgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic collapse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Palsy bells (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Transient cerebral ischemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Unilateral carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Unilateral renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteral calculus (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Ureteric calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/160 (0) | 1/148 (1) | 0/165 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/135 (0) | 0/145 (0) | 1/131 (1)
Premenopausal menorrhagia (Reproductive system and breast disorders) | 0/135 (0) | 0/145 (0) | 1/131 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Atherosclerosis generalized (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Bleeding (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mg LY2189265 (N=295) | 0.75 mg LY2189265 (N=293) | Insulin Glargine (N=296)
Abdominal pain upper (Gastrointestinal disorders) | 13 (17) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (12) | 6 (6) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 44 (62) | 34 (67) | 15 (18)
Dyspepsia (Gastrointestinal disorders) | 11 (11) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 11 (12) | 5 (5)
Heartburn (Gastrointestinal disorders) | 13 (13) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 76 (115) | 52 (74) | 9 (11)
Vomiting (Gastrointestinal disorders) | 35 (46) | 31 (49) | 5 (5)
Fatigue (General disorders) | 11 (11) | 7 (7) | 5 (6)
Oedema peripheral (General disorders) | 7 (7) | 17 (20) | 9 (9)
Bronchitis (Infections and infestations) | 7 (8) | 9 (11) | 13 (15)
Common cold (Infections and infestations) | 19 (23) | 28 (37) | 26 (33)
Flu syndrome (Infections and infestations) | 4 (6) | 9 (11) | 2 (2)
Nasopharyngitis (Infections and infestations) | 22 (27) | 1 (1) | 33 (43)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 2 (3) | 11 (12)
Urinary tract infection (Infections and infestations) | 12 (14) | 14 (16) | 11 (18)
Anorexia (Metabolism and nutrition disorders) | 11 (12) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 8 (10) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 10 (10) | 5 (5) | 5 (5)
Dyslipidemia (Metabolism and nutrition disorders) | 10 (10) | 5 (5) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 16 (21)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 13 (14) | 8 (10)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 9 (9)
Headache (Nervous system disorders) | 16 (19) | 20 (27) | 17 (20)
Hypertension (Vascular disorders) | 5 (5) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days